CLINICAL TRIAL: NCT03935048
Title: The Effect of a Higher Protein, Lower Glycemic Load Diet Containing Potato or Potato-based Products on Metabolic Health in Adults With Metabolic Syndrome
Brief Title: Diet and Health in Adults With Metabolic Syndrome
Acronym: MAPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jamie Baum, Associate Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1901172168
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Higher Protein, Low Glycemic Load with Potatoes (Experimental): Higher Protein, Low Glycemic Load with Potatoes (HPLG-P): low- to moderate- glycemic load meals containing white potatoes. Participants will consume low- to moderate-glycemic meals for 16 weeks and will need to consume at least 4 meals containing white potatoes.
  Interventions: Dietary Supplement: Higher protein, low glycemic load diet
- Higher Protein, Low Glycemic Load with Processed Potatoes (Active Comparator): Higher Protein, Low Glycemic Load with Processed Potatoes (HPLG-PP): low- to moderate- glycemic load meals containing processed white potato products. Participants will consume low- to moderate-glycemic meals for 16 weeks and will need to consume at least 4 meals containing white potatoes.
  Interventions: Dietary Supplement: Higher protein, low glycemic load diet
- Higher Protein, Low Glycemic Load - Control (Placebo Comparator): Higher Protein, Low Glycemic Load (HPLG-C): low- to moderate- glycemic load meals containing control carbohydrate (e.g. rice, pasta). Participants will consume low- to moderate-glycemic meals for 16 weeks and will need to consume at least 4 meals containing control carbohydrate sources.
  Interventions: Dietary Supplement: Higher protein, low glycemic load diet

INTERVENTIONS:
Dietary Supplement: Higher protein, low glycemic load diet — All dietary treatments will be designed to be isoenergetic within individual participants. Energy content of the diets will be individualized to ensure weight maintenance throughout the dietary intervention period using the Harris Benedict equation x 1.35. Glycemic load for the treatment groups will be calculated using the following equation:
  Glycemic Load = Glycemic Index x Grams of carbohydrates/100. Potatoes, processed potato products, and control carbohydrate foods will be provided.

SUMMARY:
The prevalence of US adults with Metabolic Syndrome (MetS) is over 34%, impacting nearly 35% of all adults and 50% of those aged 60 years or older. MetS is characterized as a combination of underlying risk factors that when, occurring together, increase the risk for chronic diseases such as type 2 diabetes mellitus (T2DM), cardiovascular disease, stroke, and certain types of cancer, resulting in an 1.6-fold increase in mortality. According the American Heart Association, health risks associated with Metabolic Syndrome can be significantly reduced by reducing body weight and eating a diet that is rich in whole grains, fruits, and vegetables. Potatoes (e.g. skin-on white potatoes) are an excellent source of potassium, vitamin C, and vitamin B6 and a good source of magnesium and dietary fiber. In addition, the potato has greater dry matter and protein per unit growing area compared with cereals. Despite this, consumers tend to believe that potatoes are high in calories and in fat compared with other carbohydrate sources such as rice or pasta, an incorrect assumption since a potato has negligible fat and a low energy density similar to legumes. Data from short-term nutrition intervention trials, suggest that potatoes consumed as part of a low-glycemic load meal can play a role in the prevention or treatment of MetS. However, the impact of long-term potato consumption on cardiometabolic risk factors associated with MetS is not known. Therefore, there is a critical need to determine if regular (> 4 times per week) potato consumption can improve cardiometabolic health in individuals with MetS.

ELIGIBILITY:
Inclusion Criteria:

* Resides in Northwest Arkansas
* Age 18+ years
* Metabolic Syndrome (characterized by participant having three or more of the following measurements: abdominal obesity, triglyceride level over 150 mg/dl, HDL cholesterol < 40 mg/dl in men and 50 mg/dl in women, systolic blood pressure of 130 mm Hg or diastolic blood pressure of 85 mm Hg, and/or fasting glucose > 100 mg/dL)
* All ethnicities
* Female and male
* Currently consuming a high glycemic load diet

Exclusion Criteria:

* Food allergies
* Dietary restrictions (e.g. vegetarian, vegan, etc.)
* Trying to lose weight in last 3 months
* Prescription medications related to heart disease or type 2 diabetes
* Fear of needles

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Serum lipid levels | Change from baseline at 16 weeks
  Total Cholesterol, LDL-Cholesterol, HDL-Cholesterol, Free Fatty Acids, Triglycerides
Plasma glucose levels | Change from baseline at 16 weeks
  Plasma glucose levels

SECONDARY OUTCOMES:
Waist circumference | Change from baseline at 16 weeks
  Waist circumference in centimeters
Dietary intake | Change of time of study (16 weeks)
  Monthly food records will be recorded to determine changes in diet intake
Mood | Change from baseline at 16 weeks
  Mood will be measured using the Profile of Mood States questionnaire
Sleep quality and duration | Change from baseline at 16 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index
Sleep duration | Change from baseline at 16 weeks
  Sleep duration will be assessed using an Actigraph sleep monitor
Marker of appetite and sleep | Change from baseline at 16 weeks
  Orexin (also known as hypocretin)
Appetite | Change from baseline at 16 weeks
  Anorexigenic appetite hormone - PYY (peptide tyrosine tyrosine)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No